CLINICAL TRIAL: NCT05341960
Title: Nourishing Beginnings: Addressing Food Insecurity Among Medicaid-Eligible Pregnant Individuals
Brief Title: Nourishing Beginnings: Addressing Food Insecurity During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Better Health Partnership (Unknown); Greater Cleveland Food Bank (Unknown); Pregnancy with Possibilities Resource Center (Unknown); Village of Healing Center (Unknown); United Way of Greater Cleveland (Unknown); MetroHealth Medical Center (Other); Cleveland Department of Public Health (Unknown)
Responsible Party: Principal Investigator, Elaine Borawski, Angela Bowen Williamson Professor of Community Nutrition, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20211072
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Related; Food Insecurity; Premature Birth; Pregnancy Complications
Keywords: Food Insecurity; Community Health Workers; Food Delivery; Prenatal Nutrition; Social Determinants of Health
MeSH Terms: conditions — Premature Birth; Pregnancy Complications | interventions — Financial Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food Delivery (Experimental): Food box delivered to participant home every 2 weeks until 6 weeks post delivery
  Interventions: Behavioral: Food Delivery
- Financial Support and Navigation (Experimental): $30 provide on gift card every two weeks until 6 weeks post delivery + neighborhood food retail navigation support.
  Interventions: Other: Financial Support
- Control Group (No Intervention): Selected from claims data, matched.

INTERVENTIONS:
Behavioral: Food Delivery — Food box with food to feed a family of four, delivered by the Greater Cleveland Food Bank every two weeks. Based on participant preferences, includes recipes.
  Arms: Food Delivery
Other: Financial Support — Provides supplemental funds to purchase healthy foods; provides choice. Includes recipes for limited budgets and assistance locating healthy food options in their specific neighborhood.
  Arms: Financial Support and Navigation

SUMMARY:
This is a pilot project designed to test the feasibility of implementing a community health worker (CHW)-led intervention to improve nutritious food access and consumption among pregnant people and to evaluate the effectiveness of this approach. The project will be conducted in partnership with the Greater Cleveland Food Bank and the Better Health Partnership Community Health Worker HUB

DETAILED DESCRIPTION:
The Nourishing Beginnings pilot study will enroll 160 pregnant individuals (<22 weeks gestation) who are eligible to use the Partnership Community HUB (i.e., Medicaid eligible). Participants will be randomly assigned into one of two intervention arms - either direct food delivery (n=80) or small financial resources and individualized navigation support for accessing local healthy foods (n=80).

The pilot will (1) assess the feasibility and allow protocol refinement; (2) assess the preliminary impact of CHW-led intervention; and (3) conduct a rigorous process evaluation of the implementation of the intervention using an effectiveness-implementation hybrid type 1 design. Dietary behavior, psychosocial health, health care utilization, and health outcomes and birth outcomes will be tracked at baseline, mid-pregnancy, and at delivery, derived from both primary and secondary data sources (i.e., Hub and claims data). Critical implementation points (referral, CHW touch points, and food delivery) will be assessed. Intervention arms will be compared to a matched comparison group derived from local claims data for the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid eligible
* Enrolls in the CHW Hub
* Able to read and understand English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Food Insecurity | Change from baseline to 10 weeks post-randomization
  6 item, United States Department of Agriculture (USDA) measure; dichotomous outcome
Food Insecurity | Change from baseline to delivery
  6 item, USDA measure; dichotomous outcome
Maternal depression | Change from baseline to 10 weeks post-randomization
  9 item, self-administered, assesses maternal depression
Maternal depression | Change from baseline to delivery
  9 item, self-administered, assesses maternal depression
Social Support | Change from baseline to 10 weeks post-randomization
  6 item, self-administered, assesses emotional and instrumental social support
Social Support | Change from baseline to delivery
  6 item, self-administered, assesses emotional and instrumental social support
Mastery | Change from baseline to 10 weeks post-randomization
  7 item, self-administered, assesses skill development and locus of control
Mastery | Change from baseline to delivery
  7 item, self-administered, assesses skill development and control
Baby Birthweight | At delivery
  Baby's birthweight, measured in grams
Baby Gestational Age | At delivery
  Baby's gestational age at birth, measured in weeks
Neonatal Intensive Care (NICU) Utilization | From date of NICU admission to date of discharge from NICU or death, which ever comes first, up to 100 months
  number of days baby was admitted to NICU
Days Hospitalization | From date of delivery to date of baby discharge from hospital or death, which ever comes first, up to 100 months
  total number of days baby was hospitalized following birth

CONTACTS AND LOCATIONS:
Overall Officials: Elaine A Borawski, PhD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Mom's First, Cleveland, Ohio
  - Better Health Partnership CHW HUB, Cleveland, Ohio

REFERENCES:
- [Derived] Borawski EA, Goodwin MA, Glenn AC, Mundorf C, Fernandez LI, Larberg N, Gunzler DD, Lever JS. Study design and protocol for Nourishing Beginnings, an integrated service delivery model addressing food insecurity and social needs of low-income pregnant individuals. Contemp Clin Trials. 2023 Oct;133:107310. doi: 10.1016/j.cct.2023.107310. Epub 2023 Aug 14. PMID 37586560

DOCUMENTS (1):
  • Informed Consent Form (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05341960/ICF_000.pdf